CLINICAL TRIAL: NCT01874353
Title: Phase III Randomised, Double Blind, Placebo Controlled Study of Olaparib Maintenance Monotherapy in Platinum Sensitive Relapsed BRCA Mutated Ovarian Cancer Patients With a Complete or Partial Response Following Platinum Based Chemotherapy
Brief Title: Olaparib Treatment in BRCA Mutated Ovarian Cancer Patients After Complete or Partial Response to Platinum Chemotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Myriad Genetic Laboratories, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0816C00002; 2013-001211-75 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Platinum Sensitive; BRCA Mutated; Relapsed Ovarian Cancer; Following Complete or Partial Response to Platinum Based Chemotherapy
Keywords: BRCA; Ovarian cancer; Chemotherapy; PARP Inhibitor; Platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib 300mg tablets (Experimental): Taken orally twice daily
  Interventions: Drug: Olaparib 300mg tablets
- Placebo tablets (Placebo Comparator): Taken orally twice daily
  Interventions: Drug: Placebo to match olaparib 300mg

INTERVENTIONS:
Drug: Olaparib 300mg tablets — 300mg Olaparib or placebo tablets taken orally twice daily until objective radiological disease progression as per RECIST as assessed by the investigator (or as long as in the investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria). Dose reduction to 250mg and subsequently 200mg is permitted following confirmation of toxicity.
  Arms: Olaparib 300mg tablets
Drug: Placebo to match olaparib 300mg — 300mg Olaparib or placebo tablets taken orally twice daily until objective radiological disease progression as per RECIST as assessed by the investigator (or as long as in the investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria). Dose reduction to 250mg and subsequently 200mg is permitted following confirmation of toxicity.
  Arms: Placebo tablets

SUMMARY:
A Phase III, randomised, double-blind, placebo-controlled, multi-centre study to assess the efficacy of olaparib maintenance monotherapy in relapsed high grade serous ovarian cancer (HGSOC) patients (including patients with primary peritoneal and / or fallopian tube cancer) or high grade endometrioid cancer with BRCA mutations (documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function)) who have responded following platinum based chemotherapy.

DETAILED DESCRIPTION:
Comparison of olaparib against a placebo in patients with ovarian cancer whose cancer has already improved by taking platinum based chemotherapy. The patients must also have a fault in their DNA which codes for the BRCA protein. The BRCA protein helps mend broken DNA in the cells of the body; if this protein doesn't work properly it can increase the chance of getting cancer. The aim of this study is to see whether patients taking olaparib tablets last longer until their cancer gets worse, compared to those taking the placebo tablet. The study is also looking to see if there is an overall improvement to how long the patients survive whilst taking olaparib tablets compared to the placebo tablets; and the quality of their life whilst living with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age.

  * Female patients with histologically diagnosed relapsed high grade serous ovarian cancer (including primary peritoneal and / or fallopian tube cancer) or high grade endometrioid cancer.
  * Documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function).
  * Patients who have received at least 2 previous lines of platinum containing therapy prior to randomisation

For the penultimate chemotherapy course prior to enrolment on the study:

• Patient defined as platinum sensitive after this treatment; defined as disease progression greater than 6 months after completion of their last dose of platinum chemotherapy

For the last chemotherapy course immediately prior to randomisation on the study:

* Patients must be, in the opinion of the investigator, in response (partial or complete radiological response), or may have no evidence of disease (if optimal cytoreductive surgery was conducted prior to chemotherapy), and no evidence of a rising CA-125, following completion of this chemotherapy course
* Patient must have received a platinum based chemotherapy regimen (e.g. carboplatin or cisplatin) and have received at least 4 cycles of treatment
* Patients must be randomized within 8 weeks of their last dose of chemotherapy
* Maintenance treatment is allowed at the end of the penultimate platinum regimen, including bevacizumab

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* BRCA 1 and/or BRCA2 mutations that are considered to be non detrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favor polymorphism" or "benign polymorphism" etc.)
* Patients who have had drainage of their ascites during the final 2 cycles of their last chemotherapy regimen prior to enrolment on the study.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Professor E Pujade-Lauraine, MD, PhD, Principal Investigator — Universite de Paris Descartes, France
Locations (126):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Palo Alto Foundation Medical Group, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Gynecologic Cancer Center, Orlando, Florida
  - North Shore University, Evanston, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson at Cooper Cancer Center, Voorhees Township, New Jersey
  - Womens Cancer Care Associates, Albany, New York
  - Winthrop Gynecologic Oncology Associates, Mineola, New York
  - OSU JamesCare at Mill Run, Hilliard, Ohio
  - Henry Joyce Cancer Clinic, Nashville, Tennessee
  - Aurora St Lukes Medical Center, Milwaukee, Wisconsin
- Australia (3):
  - Mercy Hospital for Women, Heidelberg
  - The Royal Womens Hospital, Parkville
  - Prince of Wales Hospital, Randwick
- Belgium (2):
  - U.Z. Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (10):
  - Centro Diagnóstico Barretos, Barretos
  - Centro Regional Integrado de Oncologia, Fortaleza
  - Hospital Araujo Jorge, Goiânia
  - Hospital de Caridade de Ijuí, Ijuí
  - Centro de Novos Tratamentos Itajai, Itajaí
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alagre, Porto Alegre
  - Hospital de Base São José do Rio Preto, São José do Rio Preto
  - Centro de Referencia da Saude da Mulher, São Paulo
  - Instituto do Câncer de São Paulo, São Paulo
- Canada (7):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - CHUM - Hopital Norte-Dame, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - CHUS Site Fleurimont, Sherbrooke, Quebec
- China (16):
  - Beijing Cancer Hospital, Beijing
  - The Tumor Hospital affiliated to China Medical Science Insti, Beijing
  - 1st Hospital of Jilin university, Changchun
  - Jilin Provincial Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital Affiliated to Sichuan University, Chengdu
  - ChongQing Cancer Hospital, Chongqing
  - Research Site, Guangzhou
  - Women's Hospital, Zhejaing University School of Medicine, Hangzhou
  - The Tumour Hospital of Harbin Medical University, Harbin
  - Zhejiang Cancer Hospital, Huangzhou, Huangzhou
  - JINAN, Qi Lu Hosp. of SD Univ., Jinan
  - Research Site, Shanghai
  - Shanghai Cancer Hospital of Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - First affiliated hospital college of XianJiaotong University, Xi'an
- France (12):
  - Institut Bergonie, Bordeaux
  - CAC François Baclesse, Caen
  - 69LYON, C Bérard, Onco, Lyon
  - Centre Catherine de Sienne, Nantes
  - 75PARIS, H Tenon, Onco, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Institut Curie Paris Et Saint Cloud, Paris
  - 69PIERREBE, CH Lyon Sud,, Pierre-Bénite
  - 92STCLOUD, C Huguenin, Onco, Saint-Cloud
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Helios-Kliniken Berlin - Buch, Berlin
  - Friedrich-Alexander-Universität Erlangen-Nürnberg, Erlangen
  - Klinikum Essen-Mitte,Evang. Huyssens-Stiftung/Knapps gGmbH, Essen
  - Johann-Wolfgang Goethe-Universität, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum rechts der Isar der Technischen Universität, München
  - Onkologie Ravensburg, Ravensburg
  - Universitätsklinikum Rostock, Rostock
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Sapir Medical Centre, Kfar Saba
  - Tel Hashomer, Ramat Gan
- Italy (6):
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Policlinico Di Modena, Modena
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto Irccs, Padua
  - Istituto Regina Elena-Polo Oncologico Ifo, Roma
  - Policlinico Universitario A. Gemelli, Roma
- Japan (9):
  - Hyogo Cancer Center, Akashi-shi
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka-shi
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Niigata University Medical and Dental Hospital, Niigata
  - Kindai University Hospital, Osakasayama-shi
  - Hokkaido University Hospital, Sapporo
  - Shizuoka Cancer Center, Sunto-gun
- Netherlands (4):
  - Netherlands Cancer Institute Antoni van Leeuwenhoek Hospital, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Universitair Medisch Centrum St. Radboud, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (5):
  - Niepubliczny Zaklad Opieki Zdrowotnej Innowacyjna Medycyna, Grzepnica
  - SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Onkologii Instytut im Marii Sklodowskiej-Curie, Warsaw
  - Szpital Specjalistyczny im. Swietej Rodziny SPZOZ, Warsaw
- Russia (3):
  - Chemotherapy Department, Russian Cancer Research Centre, Moscow
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - St.Petersburg City Oncology Dispensary, Dept. Gynecology, Saint Petersburg
- South Korea (4):
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (9):
  - Barcelona,H.Clinic i Provincial,Oncología, Barcelona
  - Barcelona,H.de la Sta.Creu i S.Pau,Oncología, Barcelona
  - Córdoba,H.Reina Sofía,Oncología, Córdoba
  - Gerona,H.Josep Trueta,Oncología, Girona
  - Madrid, H.C.S.Carlos,Oncología, Madrid
  - Madrid,H.12 de Octubre,Oncología, Madrid
  - Hospital Provincial de Navarra, Pamplona
  - Valencia, IVO, Oncología, Valencia
  - Valencia,H.C.U.Valencia,Oncología, Valencia
- United Kingdom (8):
  - City Hospital Birmingham Cancer Trials Team, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Arden Cancer Centre, Coventry
  - Edinburgh Cancer Research UK Centre, Edinburgh
  - Cancer Research UK and UCL Cancer Trials Centre, London
  - Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital and Institute of Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Barnicle A, Ray-Coquard I, Rouleau E, Cadoo K, Simpkins F, Aghajanian C, Leary A, Poveda A, Lheureux S, Pujade-Lauraine E, You B, Ledermann J, Matulonis U, Gourley C, Timms KM, Lai Z, Hodgson DR, Elks CE, Dearden S, Egile C, Lao-Sirieix P, Harrington EA, Brown JS. Patterns of genomic instability in > 2000 patients with ovarian cancer across six clinical trials evaluating olaparib. Genome Med. 2024 Dec 18;16(1):145. doi: 10.1186/s13073-024-01413-5. PMID 39695768
- [Derived] Frenel JS, Kim JW, Aryal N, Asher R, Berton D, Vidal L, Pautier P, Ledermann JA, Penson RT, Oza AM, Korach J, Huzarski T, Pignata S, Colombo N, Park-Simon TW, Tamura K, Sonke GS, Freimund AE, Lee CK, Pujade-Lauraine E. Efficacy of subsequent chemotherapy for patients with BRCA1/2-mutated recurrent epithelial ovarian cancer progressing on olaparib versus placebo maintenance: post-hoc analyses of the SOLO2/ENGOT Ov-21 trial. Ann Oncol. 2022 Oct;33(10):1021-1028. doi: 10.1016/j.annonc.2022.06.011. Epub 2022 Jun 27. PMID 35772665
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Poveda A, Floquet A, Ledermann JA, Asher R, Penson RT, Oza AM, Korach J, Huzarski T, Pignata S, Friedlander M, Baldoni A, Park-Simon TW, Tamura K, Sonke GS, Lisyanskaya A, Kim JH, Filho EA, Milenkova T, Lowe ES, Rowe P, Vergote I, Pujade-Lauraine E; SOLO2/ENGOT-Ov21 investigators. Olaparib tablets as maintenance therapy in patients with platinum-sensitive relapsed ovarian cancer and a BRCA1/2 mutation (SOLO2/ENGOT-Ov21): a final analysis of a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2021 May;22(5):620-631. doi: 10.1016/S1470-2045(21)00073-5. Epub 2021 Mar 18. PMID 33743851
- [Derived] Tjokrowidjaja A, Lee CK, Friedlander M, Gebski V, Gladieff L, Ledermann J, Penson R, Oza A, Korach J, Huzarski T, Manso L, Pisano C, Asher R, Lord SJ, Kim SI, Lee JY, Colombo N, Park-Simon TW, Fujiwara K, Sonke G, Vergote I, Kim JW, Pujade-Lauraine E. Concordance between CA-125 and RECIST progression in patients with germline BRCA-mutated platinum-sensitive relapsed ovarian cancer treated in the SOLO2 trial with olaparib as maintenance therapy after response to chemotherapy. Eur J Cancer. 2020 Nov;139:59-67. doi: 10.1016/j.ejca.2020.08.021. Epub 2020 Sep 23. PMID 32977221
- [Derived] Friedlander M, Gebski V, Gibbs E, Davies L, Bloomfield R, Hilpert F, Wenzel LB, Eek D, Rodrigues M, Clamp A, Penson RT, Provencher D, Korach J, Huzarski T, Vidal L, Salutari V, Scott C, Nicoletto MO, Tamura K, Espinoza D, Joly F, Pujade-Lauraine E. Health-related quality of life and patient-centred outcomes with olaparib maintenance after chemotherapy in patients with platinum-sensitive, relapsed ovarian cancer and a BRCA1/2 mutation (SOLO2/ENGOT Ov-21): a placebo-controlled, phase 3 randomised trial. Lancet Oncol. 2018 Aug;19(8):1126-1134. doi: 10.1016/S1470-2045(18)30343-7. Epub 2018 Jul 17. PMID 30026002
- [Derived] Pujade-Lauraine E, Ledermann JA, Selle F, Gebski V, Penson RT, Oza AM, Korach J, Huzarski T, Poveda A, Pignata S, Friedlander M, Colombo N, Harter P, Fujiwara K, Ray-Coquard I, Banerjee S, Liu J, Lowe ES, Bloomfield R, Pautier P; SOLO2/ENGOT-Ov21 investigators. Olaparib tablets as maintenance therapy in patients with platinum-sensitive, relapsed ovarian cancer and a BRCA1/2 mutation (SOLO2/ENGOT-Ov21): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1274-1284. doi: 10.1016/S1470-2045(17)30469-2. Epub 2017 Jul 25. PMID 28754483
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00002&attachmentIdentifier=b78b290c-58f4-42f8-902e-c6641f7cf141&fileName=d0816c00002.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global Cohort: First patient screened: 03 Sep 2013; last patient screened on 21 Nov 2014. 602 patients screened across 119 centres in 16 countries; 295 were randomized. Results are reported for analysis of PFS (DCO: 19 Sep 2016) and OS (DCO: 03 Feb 2020).
  China Cohort: First patient enrolled: 07 Apr 2015; last patient enrolled: 30 Oct 2015. 127 patients screened across 16 sites; 32 were randomized. Results are reported for analysis of PFS (DCO: 16 Jan 2017) and OS (DCO: 03 Feb 2020).
Pre-assignment Details: It was planned that approximately 264 women from the Global Cohort and 33 women from the China Cohort, with BRCA mutated relapsed ovarian cancer who are in complete or partial response following platinum based chemotherapy, were to receive olaparib 300 mg bd or matching placebo in a 2:1 ratio.
Groups:
- Olaparib 300mg Tablets (Global Cohort); Placebo Tablets (Global Cohort); Olaparib 300mg Tablets (China Cohort); Placebo Tablets (China Cohort): Taken orally twice daily
Period: Overall Study
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Started | 196 | 99 | 22 | 10
Completed | 69 | 26 | 7 | 3
Not Completed | 127 | 73 | 15 | 7
Not completed — One patient was unblinded and one patient was randomised in error | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2 | 0
Not completed — Death | 110 | 60 | 13 | 7
Not completed — Withdrawal by Subject | 13 | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Global Cohort: 196 Olaparib, 99 Placebo China Cohort: 22 Olaparib, 10 Placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300mg Tablets | Placebo Tablets | Total
Number analyzed (Participants) | 218 | 109 | 327
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: There are 196 Olaparib patients in the Global Cohort and 22 in the China Cohort (Total = 218).
  There are 99 Placebo patients in the Global Cohort and 10 in the China Cohort (Total = 109)
  Years
    Global Cohort: number analyzed (Participants) | 196 | 99 | 295
    Global Cohort | 57.0 (9.2) | 56.6 (8.9) | 56.9 (9.09)
    China Cohort: number analyzed (Participants) | 22 | 10 | 32
    China Cohort | 50.6 (8.42) | 47.4 (9.29) | 49.6 (8.68)
Age, Customized [Count of Participants; unit: Participants] — Population: There are 196 Olaparib patients in the Global Cohort and 22 in the China Cohort (Total = 218). There are 99 Placebo patients in the Global Cohort and 10 in the China Cohort (Total = 109)
  Participants
    Global Cohort: number analyzed (Participants) | 196 | 99 | 295
    Global Cohort: <50 | 38 | 25 | 63
    Global Cohort: >=50-<65 | 118 | 52 | 170
    Global Cohort: >=65 | 40 | 22 | 62
    China Cohort: number analyzed (Participants) | 22 | 10 | 32
    China Cohort: <50 | 11 | 7 | 18
    China Cohort: >=50-<65 | 10 | 2 | 12
    China Cohort: >=65 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are 196 Olaparib patients in the Global Cohort and 22 in the China Cohort (Total = 218). There are 99 Placebo patients in the Global Cohort and 10 in the China Cohort (Total = 109)
  Participants
    Global Cohort: number analyzed (Participants) | 196 | 99 | 295
    Global Cohort: Female | 196 | 99 | 295
    Global Cohort: Male | 0 | 0 | 0
    China Cohort: number analyzed (Participants) | 22 | 10 | 32
    China Cohort: Female | 22 | 10 | 32
    China Cohort: Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There are 196 Olaparib patients in the Global Cohort and 22 in the China Cohort (Total = 218). There are 99 Placebo patients in the Global Cohort and 10 in the China Cohort (Total = 109)
  Participants
    Global Cohort: number analyzed (Participants) | 196 | 99 | 295
    Global Cohort: Hispanic or Latino | 10 | 1 | 11
    Global Cohort: Not Hispanic or Latino | 186 | 98 | 284
    Global Cohort: Unknown or Not Reported | 0 | 0 | 0
    China Cohort: number analyzed (Participants) | 22 | 10 | 32
    China Cohort: Hispanic or Latino | 0 | 0 | 0
    China Cohort: Not Hispanic or Latino | 22 | 10 | 32
    China Cohort: Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: There are 196 Olaparib patients in the Global Cohort and 22 in the China Cohort (Total = 218). There are 99 Placebo patients in the Global Cohort and 10 in the China Cohort (Total = 109)
  Participants
    Global Cohort: number analyzed (Participants) | 196 | 99 | 295
    Global Cohort: WHITE | 173 | 91 | 264
    Global Cohort: BLACK OR AFRICAN AMERICAN | 1 | 0 | 1
    Global Cohort: AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0
    Global Cohort: ASIAN | 22 | 7 | 29
    Global Cohort: NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0
    Global Cohort: OTHER | 0 | 1 | 1
    China Cohort: number analyzed (Participants) | 22 | 10 | 32
    China Cohort: WHITE | 0 | 0 | 0
    China Cohort: BLACK OR AFRICAN AMERICAN | 0 | 0 | 0
    China Cohort: AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0
    China Cohort: ASIAN | 22 | 10 | 32
    China Cohort: NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0
    China Cohort: OTHER | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Using Investigator Assessment According to Modified Response Evaluation Criteria In Solid Tumours (RECIST 1.1)
Description: To determine the efficacy by progression free survival (PFS) (using investigator assessment according to modified Response Evaluation Criteria In Solid Tumours (RECIST 1.1)) of olaparib maintenance monotherapy compared to placebo in BRCA mutated relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.
Time Frame: Radiologic scans performed at baseline then every ~12 weeks up to 72 weeks, then every ~ 24 weeks thereafter until objective radiological disease progression. Assessed until 19 Sep 2016 DCO (16 Jan 2017 DCO for China Cohort); up to a maximum of 36 months.
Population: Full Analysis Set (FAS) consisting of all patients randomized as part of global enrolment, excluding China [Primary analysis] China Full Analysis Set (FAS) includes all patients who were randomised at sites in China.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | 19.1 [16.3 to 25.7] | 5.5 [5.2 to 5.8] | 13.8 [6.5 to 16.6] | 5.5 [2.7 to NA] — Insufficient PFS events to estimate upper 95% CI
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy and time to disease progression in the penultimate platinum based chemotherapy prior to enrolment; Model includes factors for response to previous platinum chemotherapy and time to disease progression in the penultimate platinum based chemotherapy; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.22 to 0.41] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes a treatment factor only; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.17 to 1.19] — A hazard ratio < 1 favours olaparib

2. Secondary Outcome: Efficacy in Patients Following Platinum Based Chemotherapy by Assessment of Overall Survival
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy by assessment of overall survival (OS).
Time Frame: Survival assessed every 4 weeks until treatment discontinues, then every 12 weeks. Assessed until 03 Feb 2020 DCO; up to a maximum of 75 months.
Population: Full Analysis Set (FAS) consisting of all patients randomized as part of global enrolment (excluding China) China Full Analysis Set (FAS) includes all patients who were randomised at sites in China.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | 51.7 [41.5 to 59.1] | 38.8 [31.4 to 48.6] | 41.7 [17.6 to NA] — Insufficient OS events to estimate upper 95% CI | 36.4 [13.2 to NA] — Insufficient OS events to estimate upper 95% CI
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p = 0.0537, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.54 to 1.00] — A hazard ratio <1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes a treatment factor only; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.38 to 2.49] — A hazard ratio <1 favours olaparib

3. Secondary Outcome: Efficacy in Patients Following Platinum Based Chemotherapy by Assessment of Time to Earliest Progression by RECIST or Cancer Antigen (CA-125) or Death
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy by assessment of time to earliest progression by RECIST or CA-125 or death.
Time Frame: CA-125 at baseline then every 4 wks. Radiologic scans at baseline then every ~12 wks up to 72 wks, then every ~ 24 wks until objective radiological disease progression. Assessed until 19Sep2016 DCO (16Jan2017 DCO for China Cohort); up to a max of 36 mths.
Population: Full Analysis Set (FAS) consisting of all patients randomized as part of global enrolment (excluding China).
  China Full Analysis Set (FAS) includes all patients who were randomised at sites in China.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | 16.9 [14.6 to 22.3] | 4.9 [3.7 to 5.6] | 12.9 [5.9 to 14.0] | 3.7 [1.0 to 7.4]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p < 0.0001, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.23 to 0.41] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes a treatment factor only; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.18 to 1.03] — A hazard ratio <1 favours olaparib

4. Secondary Outcome: Efficacy in Patients Following Platinum Based Chemotherapy by Assessment of Time From Randomization to Second Progression
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated relapsed ovarian cancer patients who are in complete response or partial response following first line platinum based chemotherapy by assessment of time from randomization up to second progression
Time Frame: Scans at baseline then every 12 wks for 72 wks, then every 24 wks until first progression. Assessments then per local practice every 12 wks until second progression. Assessed until 19Sep2016 DCO (16Jan2017 DCO for China Cohort); up to a max of 36 mths
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | NA [24.1 to NA] — Insufficient PFS2 events to estimate upper 95% CI | 18.4 [15.4 to 22.8] | NA [NA to NA] — Insufficient PFS2 events to estimate median and 95% CI | 17.3 [6.0 to 17.3]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p = 0.0002, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.34 to 0.72] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes treatment factor only; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.22 to 3.97] — A hazard ratio < 1 favours olaparib

5. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Assessed by the the Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O)
Description: To compare the effects of olaparib maintenance monotherapy compared to placebo on Health-related Quality of Life (HRQoL) as assessed by the trial outcome index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O) in BRCA mutated relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy. The TOI ranges from 0-100 and a higher score indicates a higher HRQoL.
Time Frame: Questionnaires completed by patient at baseline, Day 29 and then every 12 weeks for 12 months. Assessed until 19 Sep 2016 DCO.
Population: Full Analysis Set (FAS) consisting of all patients randomized as part of global enrolment (excluding China) with a baseline and post baseline TOI score available [This endpoint was not assessed in the China Cohort]
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in TOI over 12 months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort)
Number analyzed (Participants) | 185 | 94
Change in TOI over 12 months | -2.90 [-4.131 to -1.673] | -2.87 [-4.643 to -1.097]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p = 0.9765, Mixed Models Analysis; Fixed effects for treatment, visit and baseline TOI with the treatment by visit and baseline TOI by visit interaction. Random patient effect; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-2.191 to 2.126]

6. Secondary Outcome: Efficacy of Olaparib by Time to First Subsequent Therapy or Death (TFST)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomization to first subsequent therapy or death (TFST).
Time Frame: Time elapsed from randomization to first subsequent therapy or death. Assessed every 12 weeks following treatment discontinuation. Assessed until 03 Feb 2020 DCO; up to a maximum of 75 months.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | 27.4 [22.6 to 31.1] | 7.2 [6.3 to 8.5] | 13.9 [9.1 to 15.9] | 5.5 [1.4 to 18.4]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p < 0.0001, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.28 to 0.48] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes a treatment factor only; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.21 to 1.08] — A hazard ratio < 1 favours olaparib

7. Secondary Outcome: Efficacy of Olaparib by Time to Second Subsequent Therapy or Death (TSST)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomization to second subsequent therapy or death (TSST).
Time Frame: Time elapsed from randomization to second subsequent therapy or death. Assessed every 12 weeks following treatment discontinuation. Assessed until 03 Feb 2020 DCO; up to a maximum of 75 months.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Olaparib 300mg Tablets (ChinaCohort); Placebo Tablets (China Cohort): Taken orally twice daily
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (ChinaCohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | 35.8 [29.4 to 43.9] | 18.9 [15.5 to 21.5] | 19.0 [10.1 to 32.8] | 26.4 [6.3 to 36.0]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p < 0.0001, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.39 to 0.68] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (ChinaCohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model included treatment factor only; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.37 to 1.85] — A hazard ratio < 1 favours olaparib

8. Secondary Outcome: Efficacy of Olaparib by Time From Randomization to Study Treatment Discontinuation or Death (TDT)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomization to study treatment discontinuation or death (TDT).
Time Frame: Time elapsed from randomization to study treatment discontinuation or death. Assessed until 03 Feb 2020 DCO; up to a maximum of 75 months.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 196 | 99 | 22 | 10
Months | 19.4 [14.9 to 25.9] | 5.6 [5.0 to 6.8] | 13.4 [6.3 to 16.5] | 4.7 [1.3 to 11.1]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p < 0.0001, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.28 to 0.49] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority or Other; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes a treatment factor only; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.20 to 1.04] — A hazard ratio < 1 favours the Olaparib arm

9. Secondary Outcome: Efficacy in Patients With a Deleterious or Suspected Deleterious Variant in Either of the BRCA Genes by Assessment of PFS.
Description: To assess efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (gene sequencing and large rearrangement analysis).
Time Frame: Radiologic scans performed at baseline then every ~12 weeks for the first 72 weeks, then every ~24 weeks thereafter, assessed until disease progression. Assessed until 19 Sep 2016 DCO.
Population: Full Analysis Set (FAS) consisting of all patients randomized as part of global enrolment (excluding China) and confirmed as Myriad gBRCAm [This endpoint was not assessed in the China Cohort]
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort)
Number analyzed (Participants) | 190 | 96
Months | 19.3 [16.5 to 27.3] | 5.5 [5.0 to 5.8]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority or Other; p < 0.0001, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.22 to 0.40] — A hazard ratio < 1 favours olaparib

10. Secondary Outcome: To Determine the Exposure to Olaparib by Pharmacokinetic Analysis
Description: To determine the exposure to olaparib in patients receiving olaparib maintenance monotherapy
Time Frame: Pharmacokinetics sampling to be performed in a subset of patients. Sampling times: Day 1 pre-dose & 1 hour; Day 15 pre-dose & 1 hour; Day 29 pre-dose. Assessed until 19 Sep 2016 DCO.
Population: Pharmacokinetic (PK) Analysis Set - all patients who receive study treatment as per protocol, do not violate or deviate from the protocol in ways that would significantly affect the PK analyses and have valid PK data.
  The PK Analysis Set is a subset of the Global FAS; PK analysis was not performed in the China Cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Olaparib 300mg Tablets
Number analyzed (Participants) | 93
mcg/mL
  Day 1 - Pre-dose | NA (NA) — Prior to receiving olaparib so not calculated
  Day 1 - 1 hour | 3.26 (312.2)
  Day 15 - Pre-dose | 0.92 (95.5)
  Day 15 - 1 hour | 5.12 (61.8)
  Day 29 - Pre-dose | 0.94 (179.0)

ADVERSE EVENTS:
Time Frame: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of olaparib/placebo.
Groups:
- Olaparib 300 Tablets (Global Cohort); Placebo Tablets (Global Cohort); Olaparib 300 Tablets (China Cohort); Placebo Tablets (China Cohort): Taken orally twice daily
Arm/Group | Olaparib 300 Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300 Tablets (China Cohort) | Placebo Tablets (China Cohort)
All-Cause Mortality (participants affected / at risk) | 116/196 | 65/99 | 13/22 | 7/10
Serious Adverse Events (participants affected / at risk) | 50/195 | 8/99 | 5/22 | 1/10
Other Adverse Events (participants affected / at risk) | 192/195 | 91/99 | 21/22 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 Tablets (Global Cohort) (N=195) | Placebo Tablets (Global Cohort) (N=99) | Olaparib 300 Tablets (China Cohort) (N=22) | Placebo Tablets (China Cohort) (N=10)
Anaemia (Blood and lymphatic system disorders) | 8 (13) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 Tablets (Global Cohort) (N=195) | Placebo Tablets (Global Cohort) (N=99) | Olaparib 300 Tablets (China Cohort) (N=22) | Placebo Tablets (China Cohort) (N=10)
Anaemia (Blood and lymphatic system disorders) | 83 (149) | 9 (9) | 7 (14) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 21 (35) | 1 (1) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 27 (47) | 5 (12) | 5 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (22) | 3 (3) | 3 (5) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 13 (13) | 7 (7) | 3 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 53 (90) | 31 (34) | 3 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 24 (27) | 13 (14) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 46 (65) | 23 (30) | 1 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 67 (128) | 20 (28) | 4 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 12 (19) | 4 (4) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 10 (11) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (15) | 4 (4) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 5 (19) | 1 (5) | 2 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 20 (39) | 6 (7) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 77 (153) | 20 (27) | 8 (17) | 1 (1)
Fatigue (General disorders) | 75 (91) | 15 (22) | 7 (11) | 2 (4)
Influenza like illness (General disorders) | 15 (18) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 5 (5) | 2 (2) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 13 (14) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 4 (9) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 25 (48) | 11 (14) | 2 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (15) | 4 (4) | 3 (3) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 4 (4) | 2 (2) | 1 (3)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 20 (29) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 18 (39) | 1 (2) | 5 (12) | 1 (1)
Platelet count decreased (Investigations) | 15 (31) | 1 (1) | 4 (13) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 44 (59) | 11 (11) | 8 (10) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (23) | 7 (8) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 34 (43) | 6 (7) | 4 (4) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 29 (43) | 9 (9) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 148 (290) | 35 (48) | 18 (33) | 1 (3)
Asthenia (General disorders) | 62 (107) | 27 (29) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 13 (18) | 3 (4) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 17 (20) | 7 (8) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 28 (39) | 6 (9) | 1 (1) | 1 (2)
Cystitis (Infections and infestations) | 15 (27) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 17 (19) | 6 (6) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 11 (14) | 3 (5) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 11 (13) | 4 (6) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (25) | 6 (10) | 7 (14) | 2 (5)
Urinary tract infection (Infections and infestations) | 18 (28) | 9 (12) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
White blood cell count decreased (Investigations) | 13 (40) | 1 (2) | 5 (9) | 1 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (15) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 29 (54) | 10 (10) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (33) | 14 (14) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (43) | 13 (15) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (28) | 5 (5) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (3) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 7 (7) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (20) | 5 (8) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 38 (46) | 6 (6) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 50 (82) | 14 (15) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 11 (11) | 4 (4) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 12 (13) | 5 (5) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 14 (15) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 13 (16) | 5 (5) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 14 (20) | 9 (9) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (54) | 6 (6) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (33) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 5 (5) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (15) | 6 (6) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (16) | 5 (6) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 14 (18) | 5 (5) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The outbreak of the COVID-19 pandemic shortly before the final OS DCO (03 February 2020) was not judged to meaningfully impact the overall quality of the study, including the conduct, data, and interpretation of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days